CLINICAL TRIAL: NCT04064060
Title: A Phase 3b, Open-label, Single-arm, Rollover Study to Evaluate Long-term Safety in Subjects Who Have Participated in Other Luspatercept (ACE-536) Clinical Trials
Brief Title: A Study to Evaluate Long-term Safety in Participants Who Have Participated in Other Luspatercept (ACE-536) Clinical Trials
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-LTFU-001; U1111-1235-8123 (Registry Identifier: WHO); 2022-502498-40 (Other: EU CTR)
Record Dates: First submitted 2019-08-09; First posted 2019-08-21 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndromes (MDS); Beta-thalassemia; Myeloproliferative Neoplasm(MPN)-Associated Myelofibrosis
Keywords: ACE-536; Luspatercept; MDS; Beta-thalassemia; Myeloproliferative neoplasm (MPN)-associated myelofibrosis
MeSH Terms: conditions — Myelodysplastic Syndromes; beta-Thalassemia; Myeloproliferative Disorders | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACE-536 (Experimental): Luspatercept will be administered as a subcutaneous (SC) injection to participants by the study staff at the clinical site and administration will be documented in the subject's source record.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Luspatercept (ACE-536), an erythroid maturation agent, is a recombinant fusion protein consisting of a modified form of the extracellular domain (ECD) of the human activin receptor type IIB (ActRIIB) linked to the human immunoglobin G 1 (IgG1) Fc domain. ActRIIB receptor and its ligands are members of the transforming growth factor-β (TGF-β) superfamily. Members of the TGF-β superfamily ligands, through their binding to activin receptors, are involved in modulating the differentiation of late-stage erythrocyte precursors (normoblasts) in the bone marrow. Luspatercept for injection is formulated as a sterile, preservative-free, lyophilized cake/powder. Luspatercept for injection is available in 25 mg and 75 mg vials and when reconstituted with water for injection, each consists of 50 mg/mL luspatercept in a 10 mM citrate buffer-based solution
  Other Names: ACE-536

SUMMARY:
A Phase 3b, open-label, single-arm, rollover study to evaluate the long-term safety of luspatercept, to the following participants:

* Participants receiving luspatercept on a parent protocol at the time of their transition to the rollover study, who tolerate the protocol-prescribed regimen in the parent trial and, in the opinion of the investigator, may derive clinical benefit from continuing treatment with luspatercept
* Participants in the follow-up phase previously treated with luspatercept or placebo in the parent protocol will continue into long-term post-treatment follow-up in the rollover study until the follow-up commitments are met
* The study design is divided into the Transition Phase, Treatment Phase and Follow-up Phase. Participants will enter transition phase and depending on their background will enter either the treatment phase or the Long-term Post-treatment Follow-up (LTPTFU) phase
* Transition Phase is defined as one Enrollment visit
* Treatment Phase: For participants in luspatercept treatment the dose and schedule of luspatercept in this study will be the same as the last dose and schedule in the parent luspatercept study. This does not apply to participants that are in long-term follow-up from the parent protocol
* Follow-up Phase includes:

  - 42 Day Safety Follow-up Visit
* During the Safety Follow up, the participants will be followed for 42 days after the last dose of luspatercept, for the assessment of safety-related parameters and adverse event (AE) reporting

  - Long-term Post-treatment Follow-up (LTPTFU) Phase
* Participants will be followed for overall survival every 6 months for at least 5 years from first dose of luspatercept in the parent protocol, or 3 years of post-treatment from last dose, whichever occurs later, or until death, withdrawal of consent, study termination, or until a subject is lost to follow-up. Participants will also be monitored for progression to AML or any malignancies/pre-malignancies. New anticancer or disease related therapies should be collected at the same time schedule

Participants transitioning from a parent luspatercept study in post-treatment follow-up (safety or LTPTFU) will continue from the same equivalent point in this rollover study.

The ACE-536-LTFU-001 rollover study will be terminated, and relevant participants will discontinue from the study when all participants fulfill 5 years on the study, including treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be enrolled in this study:

1. Participant is ≥ 18 years at the time of signing the informed consent form (ICF).
2. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Participant has been participating in a luspatercept trial and continues to fulfill all the requirements of the parent protocol and the participant has been either:

   1. Assigned to luspatercept treatment, continues to receive clinical benefit in the opinion of the investigator and should continue to receive luspatercept treatment, OR
   2. Assigned to placebo arm in the parent protocol (at the time of unblinding or in follow-up) and should cross over to luspatercept treatment, OR
   3. Assigned to the Follow-up Phase of the parent protocol, previously treated with luspatercept or placebo in the parent protocol who shall continue into LTPTFU phase in the rollover study until the follow-up commitments are met (unless requirements are met as per parent protocol to crossover to luspatercept treatment).
4. Participant understands and voluntarily signs an informed consent document prior to any study-related assessments or procedures being conducted.
5. Participant demonstrates compliance, as assessed by the investigator, with the parent study protocol requirements.
6. Applies to on treatment Participants only- females of childbearing potential (FCBP) defined as a sexually mature woman who:

1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or amenorrhea due to other medical reasons does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) must:

1. Have two negative pregnancy tests as verified by the investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the participant practices true abstinence from heterosexual contact.
2. Agrees to use, and be able to comply with highly effective, contraception without interruption, 35 days prior to starting investigational product (IP), during the study therapy (including dose interruptions), and for 84 days after discontinuation of study therapy.

   7. Applies to on treatment participants only- Male participants must:

a. Agrees to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 84 days following investigational product discontinuation even if he has undergone a successful vasectomy.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Applies to on treatment participants only- Concomitant use of any medications/procedures that are prohibited in the parent luspatercept protocol.
2. Participant has met one or more criteria for study discontinuation as stipulated in the parent luspatercept protocol.
3. Applies to on treatment participants only- More than 26 days between last luspatercept dose in the parent protocol and first dose into ACE-536-LTFU-001 protocol unless dose delay or dose discontinuation criteria met.
4. Applies to on treatment participants only- Pregnant or breastfeeding females.
5. Participant has any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (eg, imprisoned or institutionalized) that would prevent the subject from participating in the study.
6. Participant has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
7. Participant has any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 42 Day Safety Follow-up Phase
  Type, frequency, severity of AEs, relationship of treatment emergent adverse events to luspatercept
Number of participants progressing to high/very high risk MDS or AML. | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
  Progression to high/very high-risk myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) (MDS and myelofibrosis [MF] only).
Percentage of participants progressing to high/very high risk MDS or AML | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
  Progression to high/very high-risk myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) (MDS and myelofibrosis [MF] only)
Number of participants developing other malignancies/pre-malignancies | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
  Development of other malignancies/pre-malignancies
Percentage of participants developing other malignancies/pre-malignancies | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
  Development of other malignancies/pre-malignancies

SECONDARY OUTCOMES:
Overall Survival | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
  Time from date of randomization until death from any cause
Number of participants developing treatment emergent extramedullary hematopoiesis (EMH) masses | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)
Percentage of participants developing treatment emergent EMH masses | Enrollment to Long-term post-treatment follow-up (Approximately, 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (143):
- United States (12):
  - Childrens Hospital Los Angeles RHU, Los Angeles, California
  - Local Institution - 971, Oakland, California
  - Local Institution - 978, Stanford, California
  - Local Institution - 975, Tampa, Florida
  - Local Institution - 970, Chicago, Illinois
  - Local Institution - 973, Boston, Massachusetts
  - Local Institution - 961, Detroit, Michigan
  - Local Institution - 969, New York, New York
  - Local Institution - 967, Cleveland, Ohio
  - Local Institution - 972, Philadelphia, Pennsylvania
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Local Institution - 100, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Local Institution - 102, Clayton, Victoria
  - Royal Prince Alfred Hospital, Camperdown
- Belgium (4):
  - Local Institution - 182, Brasschaat
  - Local Institution - 180, Bruges
  - Local Institution - 183, Ghent
  - Local Institution - 184, Leuven
- Bulgaria (2):
  - Local Institution - 220, Boulevard, Sofia
  - Local Institution - 221, Plovdiv
- Canada (3):
  - Local Institution - 262, Toronto, Ontario
  - Local Institution - 260, Toronto, Ontario
  - Local Institution - 263, Toronto, Ontario
- China (6):
  - Local Institution - 131, Beijing, Beijing Municipality
  - Local Institution - 135, Guangzhou, Guangdong
  - Local Institution - 132, Shanghai, Shanghai Municipality
  - Local Institution - 134, Chengdu, Sichuan
  - Local Institution - 130, Tianjin, Tianjin Municipality
  - Local Institution - 133, Hangzhou, Zhejiang
- France (11):
  - Local Institution - 305, Angers
  - Local Institution - 300, Créteil
  - Local Institution - 310, La Tronche
  - Local Institution - 306, Lille
  - Local Institution - 301, Marseille
  - Local Institution - 302, Paris
  - Local Institution - 307, Pessac
  - Local Institution - 304, Pierre-Bénite
  - Local Institution - 308, Strasbourg
  - Local Institution - 309, Toulouse
  - Local Institution - 303, Tours
- Germany (10):
  - Local Institution - 341, Berlin
  - Local Institution - 348, Dresden
  - Local Institution - 345, Düsseldorf
  - Local Institution - 346, Düsseldorf
  - Local Institution - 343, Halle
  - Local Institution - 342, Hamburg
  - Local Institution - 344, Hanover
  - Local Institution - 349, Leipzig
  - Local Institution - 340, Mainz
  - Local Institution - 347, München
- Greece (5):
  - Aghia Sophia' Children's General Hospital of Athens, Athens
  - Laiko General Hospital of Athens - Center of Thalassemia, Athens
  - Local Institution - 384, Athens
  - Local Institution - 383, Rio Patras
  - Local Institution - 381, Thessaloniki
- Israel (6):
  - Local Institution - 425, Afula
  - Local Institution - 420, Haifa
  - Local Institution - 422, Jerusalem
  - Local Institution - 424, Jerusalem
  - Local Institution - 421, Nahariya
  - Local Institution - 423, Petah Tikva
- Italy (20):
  - Local Institution - 478, Florence, Tuscany
  - Local Institution - 471, Florence, Tuscany
  - Local Institution - 470, Allessandria
  - Local Institution - 464, Bologna
  - Local Institution - 466, Brindisi
  - Local Institution - 477, Cagliari
  - Local Institution - 462, Ferrara
  - Ente Ospedaliero Ospedali Galliera - Centro della Microcitemia e delle Anemie Congenite, Genoa
  - Local Institution - 473, Lecce
  - Maggiore Polyclinic Hospital, IRCCS Ca' Granda, Milan
  - Local Institution - 479, Modena
  - AORN A Cardarelli, Napoli
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliero Universitaria S. Luigi Gonzaga, Orbassano
  - Local Institution - 469, Pavia
  - Local Institution - 468, Reggio Calabria
  - Local Institution - 465, Roma
  - Local Institution - 474, Rozzano
  - Local Institution - 472, Varese
  - Local Institution - 463, Verona
- Japan (16):
  - Local Institution - 610, Nagoya, Aichi-ken
  - Local Institution - 601, Kamogawa, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Japanese Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Local Institution - 605, Hitachi, Ibaraki
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Local Institution - 0979, Sendai, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Local Institution - 611, Nagasaki, Nagasaki
  - Japanese Red Cross Medical Center, Shibuya City, Tokyo
  - NTT Medical Center Tokyo, Shinagawa City, Tokyo
  - Local Institution - 612, Chiba
  - Shonan Kamakura General Hospital, Kamakura
  - Osaka Metropolitan University Hospital, Osaka
  - Local Institution - 604, Osaka
- Chronic Care Center, Hazmiyeh, Lebanon
- Malaysia (6):
  - Local Institution - 545, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Hospital Umum Sarawak, Kuching, Sarawak
- Local Institution - 580, Amsterdam, Netherlands
- Spain (8):
  - Local Institution - 681, Barakaldo
  - Local Institution - 686, Barcelona
  - Local Institution - 685, Barcelona
  - Local Institution - 687, Madrid
  - Local Institution - 682, Oviedo
  - Local Institution - 684, Salamanca
  - Local Institution - 680, Seville
  - Local Institution - 683, Valencia
- Sweden (3):
  - Local Institution - 720, Gothenburg
  - Local Institution - 722, Lund
  - Local Institution - 721, Stockholm
- Taiwan (3):
  - Local Institution - 760, Kaohsiung, San Ming Dist.
  - China Medical University Hospital, Taichung
  - Local Institution - 761, Taipei
- Thailand (3):
  - Chulalongkorn University Faculty of Medicine - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Chiang Mai University - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Tunisia (4):
  - University Hospital Farhat Hached, Sousse
  - Bone Marrow Transplant Center, Tunis
  - Aziza Othmana Hospital, Tunis
  - Military Hospital of Tunis, Tunis
- Turkey (Türkiye) (6):
  - Local Institution - 881, Adana
  - Local Institution - 885, Ankara
  - Local Institution - 882, Istanbul
  - Local Institution - 884, Istanbul
  - Local Institution - 880, Izmir
  - Local Institution - 883, Mersin
- United Kingdom (9):
  - Local Institution - 925, Aberdeen
  - Local Institution - 921, Leeds
  - Local Institution - 923, London
  - Whittington Hospital, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Local Institution - 928, London
  - Local Institution - 924, London
  - Local Institution - 929, Oxford
  - Local Institution - 926, Sutton in Ashfield

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html